CLINICAL TRIAL: NCT06250686
Title: Exercise and Nutrition Intervention in Ovarian Cancer - Development of a Care Concept and Evaluation in Routine Clinical Practice
Brief Title: Exercise and Nutrition Intervention in Ovarian Cancer
Acronym: BENITA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Charite University, Berlin, Germany (Other); University Hospital Dresden (Other); Kliniken Essen-Mitte (Other); University Hospital Tuebingen (Other); University Hospital Schleswig-Holstein (Other); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BENITA
Record Dates: First submitted 2023-12-04; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Ovarian Cancer; Malnutrition; Muscle Wasting; Fatigue
MeSH Terms: conditions — Ovarian Neoplasms; Malnutrition; Muscular Atrophy; Fatigue | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): usual care
- Intervention (Experimental): 6 month exercise and nutrition intervention
  Interventions: Behavioral: combined exercise and nutrition intervention

INTERVENTIONS:
Behavioral: combined exercise and nutrition intervention — Patients will be instructed on how to use the Physitrack app. At the start of chemotherapy, patients will be contacted by physiotherapists and dietitians from the University Medical Center Hamburg-Eppendorf either via video call using the app or by phone to discuss the first week's program. Patients can either complete the exercise program at home using the app or receive printed exercise plans in the mail to be completed with the physical therapist of their choice. The exercise program is adjusted weekly until week 9. After week 10, adjustments are made every two weeks. For each program, patients receive a 30-minute counseling session to discuss the exercises. The 30-minute nutritional counseling session occurs every two weeks. For patients receiving neoadjuvant chemotherapy, the exercise program is interrupted for the time of surgery and the two-week recovery period and resumed when chemotherapy is resumed.
  Arms: Intervention

SUMMARY:
The objective of this multicenter randomized controlled trial is to compare a 6-month exercise and nutrition intervention (intervention group, IG) aimed at maintaining or improving physical functioning and quality of life with usual care (control group, CG) in ovarian cancer patients.

The main question it aims to answer is:

• Can an exercise and nutrition program improve physical performance during and after active treatment for ovarian cancer?

Participants of the IG will undergo:

* Weeks 1-18: approximately 15-30 minutes of daily exercise (cardio, resistance, and balance exercises); nutritional counseling focusing on malnutrition (protein-energy malnutrition).
* Weeks 19-25: More intense daily training; nutritional counseling focusing on the Mediterranean diet.

The study design includes 3 survey time points:

* Baseline: After surgery and before starting chemotherapy
* T1: After chemotherapy (week 19)
* T2: After intervention (week 26)

The primary outcome is:

• 6-minute walk test, 6 months after enrollment (T2)

ELIGIBILITY:
Inclusion Criteria:

* Patients with FIGO II-IV stage ovarian, fallopian tube, or peritoneal carcinoma
* Patients must be treated with surgery and chemotherapy
* Patients receiving adjuvant or neoadjuvant chemotherapy but not yet started

Exclusion Criteria:

* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status greater than 2
* Patients with inadequate German language skills
* Patients with physical or mental impairments that make it impossible to perform the training programs or study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Test (distance in metre) | Change in the total distance from T2 (6 months after enrollment) to baseline as target
  Sub-maximal exercise test used to assess aerobic capacity and endurance

SECONDARY OUTCOMES:
6 Minute Walk Test (distance in metre) | Change in the total distance from T1 (end of chemotherapy, approx. week 18-19) to baseline as target
  Sub-maximal exercise test used to assess aerobic capacity and endurance
Global physical activity questionnaire (GPAQ) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Physical activity in minutes per day, MET minutes per week
Assessment of body composition using bioelectrical impedance analysis (BIA) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Bioelectrical impedance analyzers use an alternating electric current to measure the two components of bioelectrical impedance in the human body, resistance r and reactance Xc. In electrophysiological terms, resistance (per unit volume) correlates negatively with the amount of body fluid (body water and fat-free mass (FFM)) through which the current flows, while reactance correlates positively with the mass of body cells. The magnitude of Xc in relation to R is expressed as the phase angle (PA). From the measured R and Xc values and other subject data, additional indicators of body composition (e.g., total body water, fat-free mass, and fat mass) can be estimated using specific prediction equations based on modeling assumptions that are generally population-, age-, sex-, fat-, and disease-specific.
Grip force dynamometer | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Hand gripping force (kg)
Polyneuropathy; item derived from EORTC CIPN20 (Item 9) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Problems standing or walking, because can't longer feel the ground under feet
Patient Health Questionnaire-9 (PHQ-9) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Depression screening
Generalized Anxiety Disorder using GAD-2 | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Anxiety
Adherence to a Mediterranean diet (MEDAS) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Adherence to a Mediterranean diet is assessed using the 14-item Mediterranean Diet Adherence Screener (MEDAS).
EORTC QLQ-C30 | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Quality of life (multidimensional) across 10 subscales
EORTC OV-28 | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Quality of life (multidimensional) focusing on ovarian cancer across 7 subscales
EORT FA-12 | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Quality of life (multidimensional) focusing on fatigue
Nutritional Risk Screening (NRS 2002) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Malnutrition risk
Brief Social Support Scale (BS6) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Social support (tangible support, emotional-informational support)
Patient Activation Measure (PAM-13) | Baseline, T1: After chemotherapy (week 19), T2: (6 months after enrollment) to baseline which is after intervention (week 26))
  Patient Activation Measure

CONTACTS AND LOCATIONS:
Overall Officials: Holger Schulz, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (7):
- Germany (7):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätskrebszentrum Dresden, Dresden
  - Evang. Klinik Essen-Mitte, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum rechts der Isar der Technischen Universität München Ismaniger Straße 22, München
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No
The study protocol will be published in a peer-reviewed journal at the outset. The Statistical Analysis Plan (SAP), Informed Consent Form (ICF), and analysis code will be provided upon request, if available at the time of request.

REFERENCES:
- [Derived] Maurer T, Belau MH, Zyriax BC, Welsch G, Jagemann B, Chang-Claude J, Daubmann A, Buchholz A, Glismann K, Moeller A, Sehouli J, Woopen H, Wimberger P, Harter P, Kaiser S, Maass N, Kiechle M, Engler T, Schmalfeldt B, Schulz H. Study protocol of an exercise and nutrition intervention for ovarian cancer patients during and after first-line chemotherapy (BENITA) - a randomized controlled trial. BMC Cancer. 2024 Nov 11;24(1):1379. doi: 10.1186/s12885-024-13102-y. PMID 39528997